CLINICAL TRIAL: NCT07028853
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of Mevrometostat (PF-06821497) With Enzalutamide in Metastatic Castration-Sensitive Prostate Cancer (MEVPRO-3)
Brief Title: This Study Will Explore Whether a Combination of the Investigational Drug Mevrometostat (PF-06821497) and Enzalutamide Will Work Better Than Taking Enzalutamide Alone in Participants With mCSPC Who Are ARPI naïve.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2321008; MEVPRO-3 (Other: Alias Study Number); 2024-519369-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-04-15; First posted 2025-06-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Castration Sensitive Prostate Cancer (mCSPC); Hormone Sensitive Prostate Cancer; Prostate Cancer; Cancer of the Prostate
Keywords: Hormone Sensitive Prostate Cancer; Mevrometostat; Metastatic castration sensitive prostate cancer; PF-06821497; EZH2; enhancer of zeste homologue-2; enzalutamide; mCSPC; HSPC; Prostate cancer; castrate sensitive prostate cancer; prostatecancer-study.com; Phase 3; efficacy; safety; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PF06821497; enzalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Participants will receive mevrometostat or matching placebo in a blinded fashion. Participants, investigators and site staff, and sponsor staff will be aware that participants in both study arms are receiving enzalutamide. Enzalutamide will be provided in an open-label manner to participants in each treatment arm.
  Participants and their caregivers will be blinded to their assigned study intervention.
  Investigators and other site staff will be blinded to participants' assigned study intervention Sponsor staff will be blinded to participants' assigned study intervention, except for sponsor staff involved in the assignment or distribution of study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Participants will receive mevrometostat/PF-06821497 (875 mg) BID (twice daily) + enzalutamide 160 mg QD (once daily)
  Interventions: Drug: Mevrometostat; Drug: Enzalutamide
- Arm B (Active Comparator): Participants will receive Placebo BID (twice daily) + enzalutamide 160 mg QD (once daily)
  Interventions: Drug: Placebo; Drug: Enzalutamide

INTERVENTIONS:
Drug: Mevrometostat — Oral continuous
  Other Names: PF-06821497
  Arms: Arm A
Drug: Placebo — Oral continuous
  Arms: Arm B
Drug: Enzalutamide — Oral continuous
  Other Names: Xtandi

SUMMARY:
This study will explore whether a combination of the investigational drug mevrometostat (PF-06821497) and enzalutamide will work better than taking enzalutamide alone in participants with mCSPC who are ARPI naïve and have not yet received chemotherapy in the mCSPC setting.

DETAILED DESCRIPTION:
This is a global, multicenter, randomized, double-blind, placebo-controlled Phase 3 study evaluating mevrometostat in combination with enzalutamide versus placebo in combination with enzalutamide in participants with mCSPC who have not received systemic anticancer treatments with the exception of androgen-deprivation therapy (ADT) and first-generation antiandrogen agents. Prior therapy with up to 3 months of ADT (chemical or surgical) is allowed, with no radiographic evidence of disease progression or rising PSA levels prior to Day 1.

This study consists of a Screening Phase, Randomization, Treatment Phase, Safety Follow-up, and Long-Term Follow-up. Participants will be randomized on a 1:1 basis to receive (Arm A) mevrometostat (PF-06821497) in combination with enzalutamide, or (Arm B) placebo in combination with enzalutamide.

ELIGIBILITY:
Inclusion Criteria

* Male participants aged ≥18 years (or the minimum age of consent in accordance with local regulations) at screening.
* Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features.
* Metastatic prostate cancer documented by positive bone scan (for bone disease) or metastatic lesion(s) on CT or MRI (for soft tissue/visceral disease).
* Resolution of acute effects of any prior therapy to either baseline severity or CTCAE Grade ≤1 (except for AEs which do not constitute a safety risk in the investigator's judgement).
* Participants must have ECOG PS 0 or 1.

Exclusion Criteria

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Clinically significant cardiovascular disease.
* Known or suspected brain metastasis or active leptomeningeal disease.
* Participants must be treatment naïve at the mCSPC stage, eg, participants cannot have received any cytotoxic chemotherapy with the following exceptions: Treatment with first-generation antiandrogen (ADT) agents is allowed for mCSPC.
* Previous administration with an investigational product (drug or vaccine) within 30 days.
* Current use or anticipated need for drugs that are known strong CYP3A4/5 inhibitors and inducers (with exception of enzalutamide as part of this study).
* Inadequate organ function.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants aged ≥18 years (or the minimum age of consent in accordance with local regulations) at screening with a diagnosis of mCSPC.
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2028-09-12 (Estimated); Study Completion 2034-12-08 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | Randomization up to approximately 4 years
  rPFS is defined as the time from randomization until PD based on BICR assessment per RECIST v1.1 (soft tissue disease) and PCWG3 (bone disease), or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Randomization up to approximately 9 years
  OS defined as the time from the date of randomization until the date of death due to any cause.
Objective response in measurable soft tissue disease | Randomization up to approximately 4 years
  The proportion of participants with measurable soft tissue disease at baseline who have a confirmed objective response of CR or PR per RECIST v1.1 will be summarized along with the 95% CI.
Duration of Response (DoR) in measurable soft tissue disease | Randomization up to approximately 4 years
  The DoR is defined as the time from the first objective evidence of soft tissue response (CR or PR, whichever is earlier) to radiographic progression or death due to any cause whichever occurs first.
Prostate Specific Antigen Response | Randomization up to approximately 4 years
  The proportion of participants with a 50% decline from baseline in PSA that is confirmed by a second consecutive value at least 21 days later in participants with detectable PSA values at baseline will be calculated for each treatment arm.
Time to prostate specific antigen (PSA) progression | Randomization up to approximately 4 years
  Time from the date of randomization to the date of the first PSA progression.
Time to initiation of antineoplastic therapy | Randomization up to approximately 4 years
  Time from randomization to first use of new antineoplastic therapy for prostate cancer.
Time to first symptomatic skeletal event | Randomization up to approximately 4 years
  Time from randomization to first tumor-related symptomatic bone fracture, surgery or radiotherapy to the bone, and spinal cord compression, whichever occurs first.
Time from randomization to CRPC | Randomization up to approximately 4 years
  Time from randomization to the first date of CRPC event.
Incidence of Adverse Events | Randomization up to approximately 5 years
  Type, incidence, severity [as graded by National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) v5.0], seriousness and relationship to study medications of AEs.
To evaluate the PK of mevrometostat when dosed in combination with enzalutamide | Cycle 3 Day 1 to last PK draw at Cycle 5 Day 1 (cycle length is 28 days)
  PK characterized by pre-dose trough and post-dose plasma concentrations of PF-06821497 at selected visits.
Change from baseline in patient reported pain symptoms per Brief Pain Inventory-Short Form (BPI-SF) | Randomization up to approximately 5 years
  Analysis of Brief Pain Inventory-Short Form (BPI-SF) will be based on the pain severity score (mean of individual BPI-SF items 3, 4, 5 and 6), the pain interference score (mean of items 9A-9G), and the single BPI-SF Item 3.
Change from baseline in health-related quality of life (HRQoL) per Functional Assessment of Cancer Therapy - Prostate (FACT-P) | Randomization up to approximately 5 years
  Change from baseline in HRQoL (FACT-P total score) will be presented. The FACT-P total score will be calculated based on the participant responses to the 39 items in the FACT-P questionnaire.
Time to definitive deterioration in patient-reported health related quality of life (HRQoL) per FACT-P | Randomization up to approximately 5 years
  Defined as the time from randomization to onset of definitive deterioration in FACT-P total score, which is defined as >10 point decrease from baseline and no subsequent observations with a <10 point decrease from baseline FACT-P total score
Patient-reported outcomes in cancer specific symptoms - time to definitive deterioration | Randomization up to approximately 5 years
  Change from baseline and time to definitive deterioration in participant-reported prostate cancer specific functioning, and symptoms per EORTC QLQ-PR25
Change from baseline and time to confirmed deterioration in participant-reported fatigue symptoms per BFI | Randomization up to approximately 5 years
  Change from baseline and time to confirmed deterioration in participant-reported fatigue symptoms (fatigue severity and fatigue interference) as per BFI.
Change from baseline in participant-reported general health status per EQ-5D-5L | Randomization up to approximately 5 years
  Participants will self-rate their current state of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression by choosing 1 of 5 possible responses that record the level of severity (no problems, slight problems, moderate problems, severe problems, or extreme problems) within each dimension.
To assess circulating tumor DNA (ctDNA) at baseline and on treatment to evaluate tumor burden | Baseline up to approximately 4 years
  Evaluation of ctDNA burden at baseline and on study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (137):
- United States (45):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Goodyear, Arizona
  - Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - Highlands Oncology Group, PA, Rogers, Arkansas
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - AdventHealth Medical Group Urology of Denver, Denver, Colorado
  - Cancer Care Specialists of Illinois, Decatur, Illinois
  - Cancer Care Specialists of Illinois, O'Fallon, Illinois
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - Montefiore Medical Center- Montefiore Medical Park, The Bronx, New York
  - University Hospitals Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - TriState Urologic Services PSC Inc. dba The Urology Group, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University Hospitals Seidman Cancer Center at UH Mentor Health Center, Mentor, Ohio
  - UH Minoff Health Center at Chagrin Highlands, Orange, Ohio
  - The Centers for Advanced Urology, LLP d/b/a Keystone Urology Specialists, Lancaster, Pennsylvania
  - Grand Strand Medical Center, Myrtle Beach, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - University of Texas Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center - William P. Clements, Jr., University Hospital, Dallas, Texas
  - University of Texas Southwestern Simmons Cancer Center - Redbird, Dallas, Texas
  - University of Texas Southwestern Medical Center-Zale Lipshy University Hospital, Dallas, Texas
  - University of Texas Southwestern Simmons Cancer Center - Fort Worth, Fort Worth, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - University of Texas Southwestern Simmons Cancer Center - Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Blue Ridge Cancer Care, Blacksburg, Virginia
  - Blue Ridge Cancer Care, Low Moor, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Blue Ridge Cancer Care, Salem, Virginia
  - Blue Ridge Cancer Care, Wytheville, Virginia
  - Northwest Medical Specialties, PLLC, Bonney Lake, Washington
  - Northwest Medical Specialties, PLLC, Federal Way, Washington
  - Northwest Medical Specialties, PLLC, Gig Harbor, Washington
  - Northwest Medical Specialties, PLLC, Puyallup, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Asociación de Beneficencia Hospital Sirio Libanés, Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina
- Australia (4):
  - Orange Health Service, Orange, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Icon Cancer Centre Chermside, Chermside, Queensland
  - ICON Cancer Centre - Kurralta Park, Kurralta Park, South Australia
- UZ Leuven, Leuven, Vlaams-brabant, Belgium
- Medical Center Futuremeds, Plovdiv, Bulgaria
- Canada (8):
  - Prostate Cancer Centre, Calgary, Alberta
  - Centre of Applied Urology Research/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Centre Intégré de Santé et de Services Sociaux de la Montérégie-Centre, Greenfield Park, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Univer, Sherbrooke, Quebec
  - Diex Recherche Trois-Rivieres, Trois-Rivières, Quebec
- China (25):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Lanzhou university second hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Huai'an Hospital Affiliated to Nanjing Medical University, Huai'an, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Suining Central Hospital, Suining, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The first affiliated hospital of Ningbo university, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou
- Czechia (2):
  - Urocentrum Praha s.r.o., Prague
  - Fakultni Thomayerova nemocnice, Prague
- Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine, France
- Germany (2):
  - Urologie Neandertal - Praxis Mettmann, Mettmann, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
- Israel (7):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Yitzhak Shamir Medical Center, Ẕerifin, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Japan (14):
  - Chiba cancer center, Chiba, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - The University of Osaka Hospital, Suita, Osaka
  - Keio university hospital, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Osaka International Cancer Institute, Osaka
  - Yamagata University Hospital, Yamagata
- Tauranga Hospital, Tauranga, Bay of Plenty, New Zealand
- Poland (3):
  - Clinical Research Center Spółka z ograniczoną odpowiedzialnością MEDIC-R Sp.k, Poznan, Greater Poland Voivodeship
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow, Lesser Poland Voivodeship
  - Clinical Best Solutions Sp. z o.o. S.K., Lublin
- Privatna urologicka ambulancia, s.r.o., Trenčín, Slovakia
- South Korea (10):
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeonranamdo
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kyungpook National University Chilgok Hospital, Deagu, Taegu-kwangyǒkshi
  - Chungnam national university hospital, Junggu, Taejǒn-kwangyǒkshi
- Spain (3):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Clinico San Carlos, Madrid
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - Royal Blackburn Hospital, Blackburn, Blackburn WITH Darwen
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London, Hammersmith and Fulham
  - Maidstone Hospital, Maidstone, KENT
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2321008